CLINICAL TRIAL: NCT05106179
Title: The Efficacy and Safety of Beta-blockers Drugs in Adults With Spinal Hemangioma: a Prospective Cohort Study
Brief Title: The Efficacy and Safety of Beta-blockers Drugs in Adults With Spinal Hemangioma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Vascular Pathology, Moscow (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S_Hemangioma
Record Dates: First submitted 2021-10-18; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Spinal Tumor; Spinal Hemangioma; Beta Blocker Toxicity
Keywords: β-blockers; Vertebral Hemangioma; Efficacy
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Atenolol; Propranolol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Previously treated + Atenolol (Active Comparator): The investigators suppose the outcome might be compromised if patient has been previously treated, that's why it is going to be compared to the main cohort. The results are going to be analysed separately
  Interventions: Drug: Atenolol Pill
- Previously treated + Propranolol (Active Comparator): The investigators suppose the outcome might be compromised if patient has been previously treated, that's why it is going to be compared to the main cohort. The results are going to be analysed separately
  Interventions: Drug: Propranolol Pill

INTERVENTIONS:
Drug: Atenolol Pill — Atenolol is a second-generation hydrophilic β-1-selective adrenergic antagonist, which is primarily metabolised by the kidneys.
  Arms: Previously treated + Atenolol
Drug: Propranolol Pill — Propranolol is highly lipophilic, nonselective β-blockers, which is primarily metabolised by the liver.
  Arms: Previously treated + Propranolol

SUMMARY:
Spinal hemangioma is one of the most common benign vertebral tumours. Being mostly asymptomatic, it is still associated with a pain syndrome especially if encroaches into the neural canal.

This study is organised to evaluate the efficacy and safety of β-blockers drugs in adults with spinal hemangioma.

ELIGIBILITY:
Inclusion Criteria:

* vertebral hemangioma

Exclusion Criteria:

* symptomatic bradycardia
* AV block
* decompensated heart failure
* asthma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reducing tumor growth | 3 months
  MRI
Reducing tumor | 6 months
  MRI
Life-quality | 3 months and 6 months
  Valid questionnaires based on the ones, approved by EuroQol Organization

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Listovskaia, MD, Study Chair — The Vascular Anomalies Center (VAC) "Hemangioma",; Dmitry Romanov, MD, Study Chair — The Vascular Anomalies Center (VAC) "Hemangioma"
Locations (1):
- The Vascular Anomalies Center (VAC) "Hemangioma", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No